CLINICAL TRIAL: NCT06475196
Title: The Prospective Cohort Study of Neoadjuvant Therapy With Sintilimab (PD-1 Inhibitor) Combined With Chemotherapy in Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Prospective Cohort Study of Neoadjuvant Therapy With Sintilimab (PD-1 Inhibitor) Combined With Chemotherapy in Resectable ESCC
Status: Enrolling by invitation | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT202405-09
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Resectable Esophageal Squamous Cell Carcinoma
Keywords: neoadjuvant therapy; PD-1 inhibitor; resectable esophageal squamous cell carcinoma
MeSH Terms: interventions — sintilimab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: sintilimab combined with platinum-containing chemotherapy Q3W for 3 cycles
  Interventions: Drug: Sintilimab (PD-1 inhibitor)
- Group B: sintilimab combined with platinum-containing chemotherapy Q3W for 2 cycles + sintilimab for 1 cycle
  Interventions: Drug: Sintilimab (PD-1 inhibitor)
- Group C: sintilimab combined with platinum-containing chemotherapy for 1 cycle + sintilimab Q3W for 2 cycles
  Interventions: Drug: Sintilimab (PD-1 inhibitor)

INTERVENTIONS:
Drug: Sintilimab (PD-1 inhibitor) — to evaluate the safety and efficacy of different cycles of sintilimab in combination with platinum-containing chemotherapy as preoperative neoadjuvant therapy in patients with resectable esophageal cancer.

SUMMARY:
This study is an open-label, prospective, cohort clinical study to evaluate the safety and efficacy of different cycles of sintilimab in combination with platinum-containing chemotherapy as preoperative neoadjuvant therapy in patients with resectable esophageal cancer. In the study, all subjects who meet the enrollment criteria will be randomized 1:1:1 to receive sintilimab combined with platinum-containing chemotherapy Q3W for 3 cycles (Group A), sintilimab combined with platinum-containing chemotherapy Q3W for 2 cycles + sintilimab for 1 cycle (Group B), sintilimab combined with platinum-containing chemotherapy for 1 cycle + sintilimab Q3W for 2 cycles (Group B) as neoadjuvant therapy, and receive radical surgery within 4-6 weeks after the completion of the last neoadjuvant therapy. Whether the subjects need adjuvant therapy and adjuvant treatment regimen after surgery are determined by the investigator, and all subjects need to complete the follow-up plan formulated by the study after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative gastroscopy showed that the main body of the tumor was located.
2. Patients with potentially resectable esophageal cancer evaluated by preoperative imaging (chest contrast-enhanced CT, head CT or MRI, abdominal B-ultrasound, PET/CT), and the potentially resectable patients refer to the 2018 edition of the Diagnosis and Treatment Standards for Esophageal Cancer formulated by the National Health and Wellness Commission, defined as patients with esophageal cancer stage T2-3, N0/N+, M0 or T4a, N0-1, M0 (8th edition AJCC stage in 2017).
3. Signed informed consent and met all the inclusion criteria of this study. 4）aged 18~75 years old 5）ECOG PS score of 0-1;

Exclusion Criteria:

1. prior treatment with immune checkpoint inhibitors, including but not limited to anti-CTLA-4, anti-PD-1 and anti-PD-L1 therapeutic antibodies, and OX-40;
2. .previous systemic therapy;
3. current participation in an interventional clinical trial or receipt of another investigational drug or medical intervention within 4 weeks;
4. presence of active hemoptysis, active diverticulitis, abdominal abscess, gastrointestinal obstruction (or other factors affecting the absorption of oral medications such as inability to swallow, nausea and vomiting, abnormal physiologic function, malabsorption syndrome, etc.) that require clinical intervention
5. the presence of any signs or history of bleeding constitution; the presence of unhealed wounds, ulcers, or fractures in patients who have experienced any bleeding or hemorrhagic event ≥ CTCAE Grade 3 within 4 weeks prior to enrollment; -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an open-label, prospective, cohort clinical study to evaluate the safety and efficacy of different cycles of sintilimab in combination with platinum-containing chemotherapy as preoperative neoadjuvant therapy in patients with resectable esophageal cancer
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
complete pathologic response (pCR) | 3 mouths
  no residual tumor cells in the surgically resected tumor specimen and all sampled regional lymph nodes after neoadjuvant treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital of the Fourth Millitary Medical University, Xi'an, Shaanxi, China